CLINICAL TRIAL: NCT03579563
Title: Impact of Hearing Aid Service-delivery Model and Technology on Patient Outcomes: A Randomized Clinical Trial
Brief Title: Impact of Hearing Aid Service-delivery Model and Technology on Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Hsiang Wu (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Yu-Hsiang Wu, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201804771; 1R01DC015997-01A1 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Presbycusis
Keywords: Presbycusis; Hearing aid
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- AUD/High-end (Active Comparator): In this group, the audiologist-based fitting will be used to provide high-end hearing aids.
  Interventions: Other: AUD fitting; Device: High-end HA
- OTC+/High-end (Experimental): In this group, audiologists will provide brief services to fit high-end OTC hearing aids
  Interventions: Other: OTC+ fitting; Device: High-end HA
- OTC/High-end (Experimental): In this group, high-end OTC hearing aids will be provided to subjects.
  Interventions: Other: OTC fitting; Device: High-end HA
- AUD/Low-end (Active Comparator): In this group, the audiologist-based fitting will be used to provide low-end hearing aids.
  Interventions: Other: AUD fitting; Device: Low-end HA
- OTC+/Low-end (Experimental): In this group, audiologists will provide brief services to fit low-end OTC hearing aids.
  Interventions: Other: OTC+ fitting; Device: Low-end HA
- OTC/Low-end (Experimental): In this group, low-end OTC hearing aids will be provided to subjects.
  Interventions: Other: OTC fitting; Device: Low-end HA

INTERVENTIONS:
Other: AUD fitting — Prescription hearing aids will be fitted by audiologists using established procedures.
  Arms: AUD/High-end; AUD/Low-end
Other: OTC+ fitting — Audiology professionals provide brief services to fit preset-based OTC hearing aids, which are simulated using prescription hearing aids.
  Arms: OTC+/High-end; OTC+/Low-end
Other: OTC fitting — In this group, preset-based OTC hearing aids, which are simulated using prescription hearing aids, will be provided to subjects. Subjects will take the full initiative and responsibility for learning and using hearing aids.
  Arms: OTC/High-end; OTC/Low-end
Device: High-end HA — High-end hearing aids will be used.
  Arms: AUD/High-end; OTC+/High-end; OTC/High-end
Device: Low-end HA — Low-end hearing aids will be used.
  Arms: AUD/Low-end; OTC+/Low-end; OTC/Low-end

SUMMARY:
Age-related hearing loss is a big problem in the United States because many people have it and it affects their quality of life. Hearing aids can help, but not many people use them. One reason is that getting hearing aids can be expensive and difficult. People usually have to visit doctors, like audiologists, many times to get their hearing tested and have the hearing aids fitted and adjusted. This process is called the AUD service model in this study. Hearing aids come with different technologies and features, like directional microphones and noise reduction algorithms. These features can make hearing aids work better but also make them more expensive, which can be another barrier for people who need them.

Recently, over-the-counter (OTC) hearing aids have become available. These hearing aids are cheaper and easier to get because people can buy them directly and fit them on their own without seeing a doctor. This is called the OTC service model in this study. Another service model that could be great is a "hybrid" service model, where professionals help fit the OTC hearing aids. This hybrid model can make hearing aids both affordable and high quality.

Studies have shown that the OTC service model works as well as the AUD service model. Additionally, other research has found no big differences in how well high-end and low-end hearing aids work for patients. However, no one has studied the different service models and technology levels together in one study, and no one has looked at how well the hybrid service model (called the OTC+ service model in this study) works.

The goal of this study is to find out how the different ways of fitting hearing aids (AUD, OTC+, and OTC) and the different technology levels (high-end and low-end) affect patient outcomes. The study will take place at two sites and will be a randomized controlled trial. Participants will be randomly assigned to one of six groups, which are combinations of the three service models and two technology levels. Measurements will be taken before the hearing aids are fitted and again six to seven weeks after fitting to see how well the hearing aids are working for the patients.

DETAILED DESCRIPTION:
Age-related hearing loss presents a significant national challenge due to its high prevalence and significant quality-of-life consequences. Although hearing aids (HAs) are the primary choice for managing age-related hearing loss, their adoption rate remains low. One commonly reported reason for not adopting HAs is the financial and physical barriers associated with traditional hearing healthcare, which involves multiple visits to licensed professionals (such as audiologists) for diagnosis and a lengthy process of fitting and fine-tuning prescription HAs. This traditional service-delivery model is referred to as the AUD service model.

Additionally, a variety of technologies and features have been implemented in HAs, including multi-channel wide dynamic range compression, directional microphones, noise reduction algorithms, and wireless functionality. These technologies have evolved from basic algorithms into more sophisticated and complex designs. The high-end technologies and features often make HAs more expensive, further exacerbating the accessibility and affordability issues of traditional hearing healthcare.

In recent years, over-the-counter (OTC) HAs have emerged as an alternative to address some of the affordability and accessibility issues of the AUD service. This direct-to-consumer model enables users to self-determine hearing loss, self-fit OTC HAs, and self-manage the device without the need for professional support. This direct-to-consumer model is referred to as the OTC service model. Additionally, it has been advocated that a hybrid service model, where professionals fit OTC HAs (referred to as the OTC+ service model), could offer affordable and quality amplification interventions.

Previous clinical trials have shown that the OTC service model yields outcomes comparable to the AUD service model. Furthermore, prior research has found no statistically significant or clinically important differences in patient outcomes between high-end and low-end HAs. However, no prior research has systematically examined the effectiveness of HA fitting service models and HA technology levels in the same study. Additionally, no prior research has investigated the patient outcomes of the OTC+ service model.

The objective of the study is to determine the effect of HA fitting services (AUD, OTC+, and OTC) and technology levels (high-end and low-end) on patient outcomes. This is a two-site randomized controlled trial. Participants will be randomly assigned to one of six parallel arms, which are factorial combinations of three service models (AUD, OTC+, and OTC) and two HA technology levels (high-end and low-end). Baseline measures will be administered before HA fitting and patient outcomes will be assessed six to seven weeks post-HA fitting.

ELIGIBILITY:
Inclusion Criteria:

* adult-onset, bilateral, mild-to-moderately severe sensorineural hearing loss

  * Puretone average across 500, 1000, 2000, and 4000 Hz between 25 and 55 dB HL
  * Thresholds from 500-4000 Hz no poorer than 65 dB HL, with up to 2 thresholds outside this criterion by < 10 dB still being eligible.
* no previous hearing aid experience

Exclusion Criteria:

* Non-native speaker of English

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Wu, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from a total of 240 participants with hearing loss recruited State of Iowa, State of Tennessee and surrounding areas. The final dataset will include laboratory data (e.g., speech recognition score) and self-reported demographic and behavioral data (e.g., questionnaire). Contact the principle investigator for data access.
Time Frame: The date will be available starting 6 months after publication of the main findings of the trial.
Access Criteria: Even though the final dataset will be stripped of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of subjects with the survey data being collected. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technologies; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Abrams HB, Chisolm TH, McManus M, McArdle R. Initial-fit approach versus verified prescription: comparing self-perceived hearing aid benefit. J Am Acad Audiol. 2012 Nov-Dec;23(10):768-78. doi: 10.3766/jaaa.23.10.3. PMID 23169194
- [Background] Abrams HB, Hnath-Chisolm T, Guerreiro SM, Ritterman SI. The effects of intervention strategy on self-perception of hearing handicap. Ear Hear. 1992 Oct;13(5):371-7. doi: 10.1097/00003446-199210000-00013. PMID 1487096
- [Background] Bainbridge KE, Ramachandran V. Hearing aid use among older U.S. adults; the national health and nutrition examination survey, 2005-2006 and 2009-2010. Ear Hear. 2014 May-Jun;35(3):289-94. doi: 10.1097/01.aud.0000441036.40169.29. PMID 24521924
- [Background] Callaway SL, Punch JL. An electroacoustic analysis of over-the-counter hearing aids. Am J Audiol. 2008 Jun;17(1):14-24. doi: 10.1044/1059-0889(2008/003). PMID 18519576
- [Background] Donahue A, Dubno JR, Beck L. Guest editorial: accessible and affordable hearing health care for adults with mild to moderate hearing loss. Ear Hear. 2010 Feb;31(1):2-6. doi: 10.1097/AUD.0b013e3181cbc783. No abstract available. PMID 20040828
- [Background] Gopinath B, Schneider J, Hartley D, Teber E, McMahon CM, Leeder SR, Mitchell P. Incidence and predictors of hearing aid use and ownership among older adults with hearing loss. Ann Epidemiol. 2011 Jul;21(7):497-506. doi: 10.1016/j.annepidem.2011.03.005. Epub 2011 Apr 21. PMID 21514179
- [Background] Lin FR, Thorpe R, Gordon-Salant S, Ferrucci L. Hearing loss prevalence and risk factors among older adults in the United States. J Gerontol A Biol Sci Med Sci. 2011 May;66(5):582-90. doi: 10.1093/gerona/glr002. Epub 2011 Feb 27. PMID 21357188
- [Background] Takahashi G, Martinez CD, Beamer S, Bridges J, Noffsinger D, Sugiura K, Bratt GW, Williams DW. Subjective measures of hearing aid benefit and satisfaction in the NIDCD/VA follow-up study. J Am Acad Audiol. 2007 Apr;18(4):323-49. doi: 10.3766/jaaa.18.4.6. PMID 17580727
- [Derived] Wu YH, Stangl E, Branscome K, Oleson J, Ricketts T. Hearing Aid Service Models, Technology, and Patient Outcomes: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Jul 1;151(7):684-692. doi: 10.1001/jamaoto.2025.1008. PMID 40372746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2019 and December 2023. Participants were recruited from the an established participant registry and through mass emails to the communities around Iowa City, IA and Vanderbilt, TN.
Period: Overall Study
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Started | 49 | 45 | 52 | 45 | 46 | 53
Completed | 43 | 41 | 42 | 40 | 39 | 40
Not Completed | 6 | 4 | 10 | 5 | 7 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 4 | 1 | 2 | 3
Not completed — Health concern (unrelated to the intervention of the study) | 2 | 0 | 0 | 1 | 2 | 2
Not completed — Time/distance concern | 0 | 0 | 1 | 0 | 0 | 1
Not completed — COVID shutdown | 2 | 3 | 4 | 3 | 1 | 2
Not completed — Protocol administration error | 1 | 0 | 1 | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end | Total
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.1) | 66.7 (12.4) | 67.6 (7.4) | 67.5 (6) | 68.9 (7.3) | 69.5 (6.8) | 67.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 22 | 19 | 17 | 21 | 121
  Male | 21 | 21 | 20 | 21 | 22 | 19 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 41 | 39 | 41 | 40 | 39 | 40 | 240
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 2 | 1 | 4
  White | 41 | 38 | 42 | 39 | 37 | 37 | 234
  More than one race | 1 | 1 | 0 | 0 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hearing loss (pure-tone average) [Mean (Standard Deviation); unit: dB HL] — Hearing loss measured using pure-tone audiometer. Pure-tone average is the mean of hearing threshold at 500 Hz, 1 kHz, and 2 kHz.
  dB HL | 31.2 (7.9) | 31.8 (7.8) | 30.1 (6.8) | 31.5 (8.1) | 30.6 (7.3) | 31 (7.2) | 31 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Hearing Aid Use Measured Using In-situ Glasgow Hearing Aid Benefit Profile (EMA-GHABP-Use)
Description: The GHABP is a questionnaire that measures hearing aid (HA) users' listening experience in four situations: TV listening, small conversation in quiet, conversation in noise, and group conversation. The GHABP will be administered using smartphone-based Ecological Momentary Assessment (EMA) to collect in-situ reports. Scores from the items that evaluate patient's HA use are averaged across the four situations to form the EMA-GHABP-Use score. The score ranges from 1 (not use HA at all) to 5 (use HA all the time).
Time Frame: 7-weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | 4.4 (1.4) | 4.1 (1.6) | 3.8 (1.8) | 4.5 (1.2) | 3.8 (1.7) | 4.3 (1.5)

2. Primary Outcome: Hearing Aid Benefit Measured Using In-situ Glasgow Hearing Aid Benefit Profile (EMA-GHABP-Global)
Description: The GHABP is a questionnaire that measures hearing aid (HA) users' listening experience in four situations: TV listening, small conversation in quiet, conversation in noise, and group conversation. The GHABP will be administered using smartphone-based Ecological Momentary Assessment (EMA) to collect in-situ reports. Scores from the items that evaluate a patient's hearing disability, hearing handicap, HA benefit, and HA satisfaction are averaged across the four situations to form the EMA-GHABP-Global score. The score ranges from 1 (poorer outcome) to 5 (better outcome).
Time Frame: 7-weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | 4.1 (.5) | 3.9 (0.6) | 3.9 (0.6) | 4.1 (0.5) | 3.8 (0.6) | 3.9 (0.5)

3. Secondary Outcome: Change of Hearing Aid Performance Measured Using the Profile of Hearing Aid Performance (PHAP)
Description: The PHAP is a questionnaire designed to measures the performance of hearing aids in speech communication. The score ranges from 1 (good performance) to 99 (poor performance) (i.e., lower scores mean better performance). Participants will complete this questionnaire pre-intervention and at 7 weeks post-intervention. The change in scores between pre- and post-intervention will be used for analysis, with score changes ranging from -98 (indicating a benefit from hearing aids) to +98 (indicating a detrimental effect of hearing aids).
Time Frame: pre-intervention and 7 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | -17.7 (20.1) | -14.2 (11.2) | -15.2 (19.7) | -16.1 (12.3) | -13.4 (14.2) | -13.6 (14.3)

4. Secondary Outcome: Change of Speech Recognition Performance as Measured by the Connected Speech Test (CST)
Description: The CST is a speech recognition test designed to simulate daily speech communication. The score ranges from 0 (understand no speech) to 100 (understand all speech). Participants will complete this questionnaire pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention will be used for analysis, with score changes ranging from -100 (indicating a detrimental effect of hearing aids) to +100 (indicating a benefit from hearing aids).
Time Frame: pre-intervention and 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: percentage of correct response
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
percentage of correct response | 10.5 (15.7) | 5 (12.4) | 6.7 (11.6) | 4.6 (10.7) | 2.2 (12.9) | 6.4 (19.7)

5. Secondary Outcome: Change of Hearing Handicap Measured by Hearing Handicap Inventory for the Elderly (HHIE) or Hearing Handicap Inventory for Adults (HHIA)
Description: The HHIE and HHIA are questionnaires designed to measure subject's perceived hearing handicap. For subjects order and younger 65 years old, the HHIE and HHIA will be used, respectively. The score ranges from 0 (no handicap) to 100 (more handicap) (i.e., lower scores mean less handicap). Participants will complete this questionnaire pre-intervention and at 7 weeks post-intervention. The change in scores between pre- and post-intervention will be used for analysis, with score changes ranging from -100 (indicating a benefit from hearing aids) to +100 (indicating a detrimental effect of hearing aids).
Time Frame: pre-intervention and 7 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | -23.3 (24.6) | -13.7 (16.6) | -15 (14.8) | -17.7 (14.9) | -14 (18.6) | -13 (17.4)

6. Secondary Outcome: Hearing Aid Use Measured Using Retrospective Glasgow Hearing Aid Benefit Profile (Retro-GHABP-Use)
Description: The GHABP is a questionnaire that measures hearing aid (HA) users' listening experience in four situations: TV listening, small conversation in quiet, conversation in noise, and group conversation. The GHABP will be administered using retrospective questionnaires. Scores from the items that evaluate patient's HA use are averaged across the four situations to form the Retro-GHABP-Use score. The score ranges from 1 (not use HA at all) to 5 (use HA all the time).
Time Frame: 6-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | 4.3 (0.9) | 3.9 (1) | 3.5 (1.2) | 4.2 (0.8) | 3.4 (1.1) | 4 (0.9)

7. Secondary Outcome: Hearing Aid Benefit Measured Using Retrospective Glasgow Hearing Aid Benefit Profile (Retro-GHABP-Global)
Description: The GHABP is a questionnaire that measures hearing aid (HA) users' listening experience in four situations: TV listening, small conversation in quiet, conversation in noise, and group conversation. The GHABP will be administered using retrospective questionnaires. Scores from the items that evaluate a patient's hearing disability, hearing handicap, HA benefit, and HA satisfaction are averaged across the four situations to form the Retro-GHABP-Global score. The score ranges from 1 (poorer outcome) to 5 (better outcome).
Time Frame: 6 weeks post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | 3.9 (0.5) | 3.7 (0.5) | 3.7 (0.5) | 3.9 (0.5) | 3.5 (0.7) | 3.7 (0.5)

8. Secondary Outcome: Hearing Aid Satisfaction as Measured by the Satisfaction With Amplification in Daily Life (SADL)
Description: The SADL is a questionnaire designed to measures subject's perceived hearing aid satisfaction. The score ranges from 1 (low satisfaction) to 7 (high satisfaction).
Time Frame: 7-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
Number analyzed (Participants) | 43 | 41 | 42 | 40 | 39 | 40
score on a scale | 5.4 (0.9) | 4.9 (1) | 4.9 (0.8) | 5.4 (0.8) | 4.8 (1) | 4.7 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject during their participation in the study, which averaged 7weeks from the time the participants entered the study.
Arm/Group | AUD/High-end | OTC+/High-end | OTC/High-end | AUD/Low-end | OTC+/Low-end | OTC/Low-end
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41 | 0/42 | 0/40 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/42 | 0/40 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/42 | 0/40 | 0/39 | 0/40

LIMITATIONS AND CAVEATS:
Firstly, the study used only one preset-based over-the-counter (OTC) device by simulation, which may not capture the variability and range of OTC hearing aids available on the market. Additionally, because participants were randomly assigned to intervention groups in the study, our OTC participants may not represent real-world users who actively choose OTC hearing aids. These limitations could affect the generalizability of study's findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03579563/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03579563/ICF_002.pdf